CLINICAL TRIAL: NCT04752644
Title: A Phase 2a, Randomised, Double-Blinded, Placebo-Controlled Study to Assess the Safety, Immunogenicity and Efficacy of the Recombinant MVA-BN®-RSV Vaccine Against Respiratory Syncytial Virus Infection in the Virus Challenge Model in Healthy Adult Participants
Brief Title: Phase 2a Study of MVA-BN-RSV Vaccination and RSV Challenge in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RSV-MVA-015
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: RSV Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group1: MVA-BN-RSV (Experimental): Participants will receive one intramuscular injection of MVA-BN-RSV (nominal titre 5 x 10*8 Inf.U per 0.5 mL) given on day -28 before RSV challenge on day 0.
  On day 0, intranasal challenge with RSV-A (Memphis 37b strain) virus will occur for all participants
  Interventions: Biological: MVA-mBN294B
- Group 2: Placebo (Placebo Comparator): Participants will receive one intramuscular injection of Tris-Buffered-Saline (0.5 mL) given on day -28 before RSV challenge on day 0.
  On day 0, intranasal challenge with RSV-A (Memphis 37b strain) virus will occur for all participants
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: MVA-mBN294B — MVA-BN-RSV (nominal titre 5 x10*8 Inf.U per 0.5 mL) as intramuscular injections. Liquid frozen suspension, single dose of 0.5ml.
  Arms: Group1: MVA-BN-RSV
Drug: Placebo — TBS (Placebo) as intramuscular injections (0.5ml)
  Arms: Group 2: Placebo

SUMMARY:
A Phase 2a, Randomised, Double-Blinded, Placebo-Controlled Study to Assess the Safety, Immunogenicity and Efficacy of the Recombinant MVA-BN®-RSV Vaccine against Respiratory Syncytial Virus Infection in the Virus Challenge Model in Healthy Adult Participants

ELIGIBILITY:
Inclusion Criteria:

1. An informed consent document signed and dated by the participant and the Investigator 2. Aged between 18 and 50 years old on the day of signing the consent form 3. In good health with no history, or current evidence, of clinically significant medical conditions, and no clinically significant test abnormalities that will interfere with participant safety, as defined by medical history, physical examination, (including vital signs), ECG, and routine laboratory tests as determined by the Investigator 4. A documented medical history prior to enrolment 5. The following criteria are applicable to female participants participating in the study.

1. Females of childbearing potential must have a negative pregnancy test prior to enrolment.
2. Females of non-childbearing potential:
3. Post-menopausal* females; defined as having a history of amenorrhea for >12 months with no alternative medical cause, and /or by FSH level >40mLU/mL, confirmed by laboratory.
4. Documented status as being surgically sterile (hysterectomy, bilateral salpingectomy and bilateral oophorectomyhysterectomy, bilateral salpingectomy and bilateral oophorectomy) 6. The following criteria apply to female and male participants:

a. Female participants of childbearing potential must use one form of highly effective contraception. Hormonal methods must be in place from at least 2 weeks prior to the first study visit. The contraception use must continue until 28 days after the date of viral challenge. Highly effective contraception is as described below: i. Established use of hormonal methods of contraception described below (for a minimum of 2 weeks prior to the first study visit). When hormonal methods of contraception are used, male are required to use a condom with a spermicide: ii. combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

1. oral 2. intravaginal 3. transdermal iii. progestogen-only hormonal contraception associated with inhibition of ovulation:

1. oral
2. injectable
3. implantable iv. Intrauterine device (IUD) v. Intrauterine hormone-releasing system (IUS) vi. Bilateral tubal ligation vii. Male sterilisation (with the appropriate post vasectomy documentation of the absence of sperm in the ejaculate) where the vasectomised male is the sole partner for that woman.

   viii. True abstinence - sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the participant.

   b. Male participants must agree to the contraceptive requirements below from the vaccination visit and continue until 28 days after the date of Viral challenge: i. Use a condom with a spermicide to prevent pregnancy in a female partner or to prevent exposure of any partner (male and female) to the IMP.

   ii. Male sterilisation with the appropriate post vasectomy documentation of the absence of sperm in the ejaculate (please note that the use of condom with spermicide will still be required to prevent partner exposure). This applies only to males participating in the study.

   iii. In addition, for female partners of childbearing potential, that partner must use another form of contraception such as one of the highly effective methods mentioned above for female participants.

   i. True abstinence - sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the participant.

   c. In addition to the contraceptive requirements above, male participants must agree not to donate sperm following discharge from Quarantine until 28 days after the date of Viral Challenge/last dosing with IMP (whichever occurs last).

7. Sero-suitable to the challenge virus, as defined in the study Analytical Plan.

Exclusion Criteria:

1. History of, or currently active, symptoms or signs suggestive of upper or lower respiratory tract infection within 4 weeks prior to the first study visit
2. Any history or evidence of any other clinically significant or currently active systemic comorbidities including psychiatric disorders (includes participants with a history of depression and/or anxiety).
3. And/or other major disease that, in the opinion of the Investigator, may put the participant at undue risk, or interfere with a participant completing the study and necessary investigations (e.g autoimmune disease or immunodeficiency).
4. Participants who have smoked ≥10 pack years at any time [10 pack years is equivalent to one pack of 20 cigarettes a day for 10 years].
5. A total body weight ≤50 kg or Body Mass Index (BMI) ≤18 kg/m2 or ≥35kg/m2.
6. Females who:

   1. Are breastfeeding, or
   2. Have been pregnant within 6 months prior to the study.
7. History of anaphylaxis-and/or a history of severe allergic reaction or significant intolerance to any food or drug or vaccine, as assessed by the PI.
8. Venous access deemed inadequate for the phlebotomy and cannulation demands of the study
9. Any significant abnormality altering the anatomy of the nose in a substantial way or nasopharynx that may interfere with the aims of the study and in particular any of the nasal assessments or viral challenge, (historical nasal polyps can be included, but large nasal polyps causing current and significant symptoms and/or requiring regular treatments in the last month will be excluded).
10. Any clinically significant history of epistaxis (large nosebleeds) within the last 3 months of the first study visit and/or history of being hospitalized due to epistaxis on any previous occasion.
11. Any nasal or sinus surgery within 3 months of the first study visit.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Area under the viral load-time curve (VL-AUC) of RSV-A Memphis 37b | From Day 2 post-viral challenge up to discharge from Quarantine (Day12).
  Median VL-AUC of RSV-A Memphis 37b as determined by qRT-PCR from nasal washes collected twice daily

SECONDARY OUTCOMES:
Peak viral load of RSV-A Memphis 37b | From Day 2 post-viral challenge up to discharge from Quarantine (Day12).
  Peak viral load of RSV-A Memphis 37b is defined by the maximum viral load in nasal washes
Total clinical symptom score (TSS) | From Day 1 post-viral challenge up to discharge from Quarantine (Day12).
  Total clinical symptom score (TSS) determined as the sum of the scores as collected on the participants' symptom diary cards, collected three times daily.
Percentage of participants with RT-PCR-confirmed RSV infection | From Day 2 up to discharge from Quarantine (Day12)
  RT-PCR-confirmed RSV infection [at least two detectable (≥LLOD) qRT-PCR measurements (reported on 2 or more consecutive days), starting two days post-viral challenge (Day 2) up to discharge from Quarantine], AND 1 or more positive clinical symptoms of Grade 2 or more from any category in the symptom scoring system (Upper Respiratory, Lower Respiratory, Systemic)
Weight of mucus produced | From Day 1 post-viral challenge up to discharge from Quarantine (Day12).
  Median AUC of mucus weight produced
Occurrence of solicited local reactions and systemic events | From day of vaccination (Day-28) and 7 subsequent days) after vaccination
  Local reactions (pain, swelling, redness, induration, itching) and systemic events (including body temperature)
Occurrence of unsolicited adverse events (AEs) | Between vaccination (Day-28) and inoculation with RSV Memphis 37b (Day0)
  Unsolicited AEs are defined as AEs observed by the participant or investigator which are not pre-listed on the memory aid card/symptom score card
Occurrence of medically attended AEs (MAEs) | From vaccination (Day -28) up to study end (Day 155 (±14 days)).
  A medically attended adverse event (MAE) is an adverse event, whether considered related to the investigational vaccine or not, that led to the participant seeking evaluation by a healthcare provider
Serious adverse events (SAEs) | From vaccination (Day -28) up to study end (Day 155 (±14 days)).
  SAEs are defined as any untoward medical occurrence that at any dose:
  results in death, is life threatening, required inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, is an important medical event
Occurrence of unsolicited AEs | From Day 0 up to Day 28 follow up
  Unsolicited AEs are defined as AEs observed by the participant or investigator which are not pre-listed on the memory aid card/symptom score card
Occurrence of SAEs | From Day 0 up to Day 28 follow up
  Occurrence of SAEs related to the viral challenge

CONTACTS AND LOCATIONS:
Locations (1):
- hVIVO Services Limited, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jordan E, Kabir G, Schultz S, Silbernagl G, Schmidt D, Jenkins VA, Weidenthaler H, Stroukova D, Martin BK, De Moerlooze L. Reduced Respiratory Syncytial Virus Load, Symptoms, and Infections: A Human Challenge Trial of MVA-BN-RSV Vaccine. J Infect Dis. 2023 Oct 18;228(8):999-1011. doi: 10.1093/infdis/jiad108. PMID 37079393